CLINICAL TRIAL: NCT06334172
Title: The Role of Oxytocin in Regulating Blood Glucose
Acronym: GLOXY-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-23071221
Record Dates: First submitted 2024-03-08; First posted 2024-03-27 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Glucose Metabolism Disorders (Including Diabetes Mellitus)
Keywords: oxytocin; blood glucose; glucose stabilization
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, single-arm study. Each participant goes through three experimental days in a randomized order - acting as their own controls
Who Masked: Participant, Investigator
Masking Description: The randomized order of infusions is blinded to both participant and investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Infusion of placebo
  Interventions: Other: Placebo
- Oxytocin 0.1 IU/min (Experimental): Infusion of oxytocin 0.1 IU/min
  Interventions: Drug: Oxytocin
- Oxytocin 0.2 IU/min (Experimental): Infusion of oxytocin 0.2 IU/min
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin
  Arms: Oxytocin 0.1 IU/min; Oxytocin 0.2 IU/min
Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
Investigating the effect of oxytocin on pancreatic endocrine functions by determining insulin and glucagon secretion within physiological ranges of plasma glucose.

DETAILED DESCRIPTION:
Insulinotropic effects of oxytocin will be examined in 20 healthy men with body mass index (BMI) < 27 kg/m2, during a graded glucose infusion test with concomitant intravenous infusion of synthetic oxytocin or placebo in a randomized, double-blinded design. This will determine the effect of oxytocin on glucose-stimulated insulin and glucagon secretion. Additional changes in plasma/serum concentrations of C-peptide, glucose, glucose-dependent insulinotropic polypeptid (GIP), glucagon-like peptide 1 (GLP-1), and lipids will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-25 kg/m2

Exclusion Criteria:

* Diabetes
* Heart-, liver or kidney disease
* More than 14 units of alcohol weekly, or drug abuse
* Smoking or any kind of nicotine products
* Alanin aminotransferase (ALAT) ≥ 2 × normal range
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1,73m2 or creatinine above normal range
* Blood pressure > 140/90
* Hemoglobin < normal range
* Corrected QT Interval (Qtc) >0,45 sec. at electrocardiogram (ECG) at screening
* Known disease in the pituitary gland or previous pituitary surgery
* Any other disease/condition which the trial managers believe may affect participation in the trial

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin secretion - c-peptide | From time 0 to time 180 min
  Insulin secretion, measured as percentual increase of area under the curve (AUC) for circulating c-peptide

SECONDARY OUTCOMES:
Glucose | From time 0 minutes to time 180 minutes
  measured as percentual increase of AUC for circulating levels
Insulin | From time 0 minutes to time 180 minutes
  measured as percentual increase of AUC for circulating levels
Glucagon | From time 0 minutes to time 180 minutes
  measured as percentual increase of AUC for circulating levels
GIP | From time 0 minutes to time 180 minutes
  measured as percentual increase of AUC for circulating levels
GLP-1 | From time 0 minutes to time 180 minutes
  measured as percentual increase of AUC for circulating levels
Lipids | From time 0 minutes to time 180 minutes
  measured as percentual increase of AUCfor circulating levels
Cross-linked C-telopeptide of type I collagen( CTX) | From time 0 minutes to time 180 minutes
  measured as percentual increase of AUC for circulating levels
Procollagen type I N-terminal propeptide (P1NP) | From time 0 minutes to time 180 minutes
  measured as percentual increase of AUC for circulating levels

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All published data will be made available to other researchers upon reasonable request